CLINICAL TRIAL: NCT07023029
Title: A Study to Assess the Effect of Etavopivat on Cardiac Repolarisation in Healthy Participants
Brief Title: A Study on the Effect of Etavopivat on Heart Rhythm in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN7535-7975; U1111-1314-5780 (Other: Universal Trial Number)
Record Dates: First submitted 2025-06-08; First posted 2025-06-15 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers; Sickle Cell Disease; Thalassemia
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A- Etavopivat (Experimental): Participants will receive a single dose of etavopivat.
  Interventions: Drug: Etavopivat
- Part A- Placebo (Placebo Comparator): Participants will receive a single dose of placebo.
  Interventions: Drug: Placebo
- Part B- Etavopivat (Experimental): Participants will receive a single dose of etavopivat.
  Interventions: Drug: Etavopivat
- Part B- Moxifloxacin (Other): Participants will receive a single dose of moxifloxacin.
  Interventions: Drug: Moxifloxacin
- Part B- Placebo (Placebo Comparator): Participants will receive a single dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etavopivat — Etavopivat will be administered orally.
  Arms: Part A- Etavopivat; Part B- Etavopivat
Drug: Moxifloxacin — Moxifloxacin will be administered orally.
  Arms: Part B- Moxifloxacin
Drug: Placebo — Placebo matching Etavopivat will be administered orally.
  Arms: Part A- Placebo; Part B- Placebo

SUMMARY:
Novo Nordisk is developing a new study medicine, Etavopivat, to treat individuals with sickle cell disease (SCD). The purpose of the study is to determine the effect of Etavopivat on the electrical activity of the heart in healthy participants. The study comprises two parts: Part A and Part B. Part A investigates the safety of a high dose of Etavopivat. In this phase, participants will receive either a single dose of Etavopivat or a placebo. Which treatment the participant gets is decided by chance. In Part B, participants will get four different treatments on four different occasions: Etavopivat in 2 different doses (the new medicine that cannot be prescribed), a dummy medicine (placebo), and an already approved medicine (moxifloxacin). The order of the 4 study medicines is decided by chance. There will be a break of 7 days between each treatment. For Part A, the study duration will be from 10 to 36 days, and for Part B, the study duration will be from 27 to 53 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Aged 18-55 years (both inclusive) at the time of signing informed consent.
* Body mass index (BMI) between 18.0 and 32.0 kilograms per square meter (kg/m^2) (both inclusive) at screening.
* Body weight above 40.0 kg at screening.
* Considered to be generally healthy based on the medical history, physical examination and the results of vital signs, electrocardiogram (ECG) and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using adequate contraceptive methods, as defined in Appendix 4, Section 10.4.
* Current participation (i.e., signed informed consent) in any other interventional clinical study.
* Exposure to an investigational medicinal product within 30 days or 5 half-lives of the investigational medicinal product (IMP) (if known), whichever is longer, before screening.
* Any condition which in the investigator's opinion might jeopardise the participant's safety or compliance with the protocol.
* Second or 3rd degree atrioventricular-block, prolongation of the QRS complex over 120 milliseconds (ms)., or of the corrected QT interval using the Fredericia formula (QTcF) over 450 ms for males and 470 ms for females, prominent U waves, or any other clinically significant abnormal ECG results or changes that make ECGs unsuitable for QT evaluations as judged by the investigator, at screening.
* Use of tobacco and nicotine products, defined as any of the below:
* Has used any product containing tobacco or nicotine within 90 days prior to screening.
* Unable or unwilling to refrain from the use of any product containing tobacco or nicotine throughout the study.
* Positive nicotine test at screening.
* Participant is unable to refrain from or anticipates the use of antacids, iron, or any drug known to be a moderate or strong inhibitor or inducer of uridine 5'-diphosphoglucuronosyltransferase (UGT) enzymes, cytochrome P450 (CYP) 3A4, CYP2C9 or permeability glycoprotein (P-gp), including St. John's Wort, for 28 days prior to dosing and throughout the study (Section 6.8).
* Participant is unable to refrain from or anticipate the use of any medications or substances prohibited in the study (Sections 5.3, 5.5 and 6.8).

A minimum of 20% African-American participants will be included in each part of this study.

Efforts will be made to include at least 40 percentage (%) of each sex into each part of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2025-06-09 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Part A: Number of treatment-emergent adverse events (AEs) | From dosing (Day 1) until end of study (Day 8)
  Measured as count of events.
Part B: Change from baseline in Fridericia heart rate corrected QT interval (ΔQTcF) for etavopivat | From pre-dose to post etavopivat/ etavopivat placebo dose on day 1 to day 23
  Measured as milliseconds.

SECONDARY OUTCOMES:
Part A: Number of treatment-emergent clinically significant abnormal findings in electrocardiogram (ECGs) | From dosing (Day 1) until end of study (Day 8)
  Measured as count of treatment-emergent clinically significant abnormal findings in ECGs.
Parts A and B: Cmax,etavopivat- Maximum observed etavopivat plasma concentration after a single dose | Day 1 (Part B)/ From day 1 to day 5 (Part A) after investigational medicinal product (IMP) administration
  Measured as nanograms per milliliter (ng/mL).
Parts A and B: AUC0-last,etavopivat- Area under the etavopivat plasma concentration-time curve from 0 hours to the time of last quantifiable concentration | Day 1 (Part B)/ From day 1 to day 5 (Part A) after IMP administration
  Measured as hours*nanograms per milliliter (h*ng/mL).
Parts A and B: AUC0-inf,etavopivat- Area under the etavopivat plasma concentration-time curve from 0 hours and extrapolated to infinity after a single dose | Day 1 (Part B)/ From day 1 to day 5 (Part A) after IMP administration
  Measured as h*ng/mL.
Parts A and B: tmax,etavopivat- Time to maximum observed etavopivat plasma concentration after a single dose | Day 1 (Part B)/ From day 1 to day 5 (Part A) after IMP administration
  Measured as hours.
Parts A and B: t½ etavopivat- Terminal half-life for etavopivat after a single dose | Day 1 (Part B)/ From day 1 to day 5 (Part A) after IMP administration
  Measured as hours.
Parts A and B: CL/F etavopivat- Apparent plasma clearance of etavopivat after a single dose | Day 1 (Part B)/ From day 1 to day 5 (Part A) after IMP administration
  Measured as liters per hour (L/h).
Parts A and B: Vz/F etavopivat- Apparent volume of distribution of etavopivat after a single dose based on plasma concentration values | Day 1 (Part B)/ From day 1 to day 5 (Part A) after IMP administration
  Measured as liters (L).
Part B: ΔQTcF for moxifloxacin | From pre-dose to post moxifloxacin dose on day 1 to day 23
  Measured as milliseconds.
Part B: Change from baseline in heart rate (ΔHR). Categorical outliers for HR | From pre-dose to post etavopivat/ etavopivat placebo dose on day 1 to day 23
  Measured as milliseconds.
Part B: Change from baseline in PR interval (ΔPR). Categorical outliers for PR | From pre-dose to post etavopivat/ etavopivat placebo dose on day 1 to day 23
  Measured as milliseconds.
Part B: Change from baseline in QRS complex duration (ΔQRS). Categorical outliers for QRS | From pre-dose to post etavopivat/ etavopivat placebo dose on day 1 to day 23
  Measured as milliseconds.
Part B: Frequency of treatment emergent changes of ECG morphology | From pre-dose to post etavopivat/ etavopivat placebo dose on day 1 to day 23
  Measured as count of treatment emergent changes of ECG morphology.
Part B: Change from baseline in ΔHR. Categorical outliers for HR | From pre-dose to post moxifloxacin dose on day 1 to day 23
  Measured as milliseconds.
Part B: Change from baseline in ΔPR. Categorical outliers for PR | From pre-dose to post moxifloxacin dose on day 1 to day 23
  Measured as milliseconds.
Part B: Change from baseline in ΔQRS. Categorical outliers for QRS | From pre-dose to post moxifloxacin dose on day 1 to day 23
  Measured as milliseconds.
Part B: Frequency of treatment emergent changes of ECG morphology | From pre-dose to post moxifloxacin dose on day 1 to day 23
  Measured as count of treatment emergent changes of ECG morphology.
Part B: ΔQTcF for etavopivat | From pre-dose to post etavopivat/etavopivat placebo dose on day 1 to day 23
  Measured as milliseconds.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- PAREXEL Intl - EPCU-Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com